CLINICAL TRIAL: NCT02581917
Title: A Study of the Metabolic Changes in Leukemia Cells Following Treatment in AML Patients
Brief Title: Metabolic Changes in Blood Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00034202; NCI-2015-01267 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 22A15 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2015-08-10; First posted 2015-10-21 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (metabolic changes): Patients undergo collection of PBMC samples for analysis via cell isolation, glycolytic flux and oxygen consumption assays, viability assays, and western blot at baseline, 24, 48, and 72 hours after starting chemotherapy.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo collection of PBMC samples
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Undergo metabolic analysis

SUMMARY:
This research trial studies metabolic changes in blood samples from patients with acute myeloid leukemia. Studying samples of blood from patients with acute myeloid leukemia in the laboratory may help doctors learn more about cancer and the development of drug resistance.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the metabolic adaptations that occur following exposure to standard chemotherapeutic agents using peripheral blood mononuclear cells from acute myeloid leukemia (AML) patients.

OUTLINE:

Patients undergo collection of peripheral blood mononuclear cell (PBMC) samples for analysis via cell isolation, glycolytic flux and oxygen consumption assays, viability assays, and western blot at baseline, 24, 48, and 72 hours after starting chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to initiate chemotherapy for either an initial diagnosis of AML or relapsed AML
* Starting the initial induction phase of therapy
* Exposure to hydroxyurea is acceptable but must be noted at the time of sample collection
* Ability to understand and the willingness to sign an institutional review board (IRB)-approved informed consent

Exclusion Criteria:

* Received at least one dose of chemotherapy during the current cycle (excluding hydroxyurea).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Acute Myeloid Leukemia (AML)
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Glycolytic flux rate | Up to 72 hours after starting chemotherapy
  Results will be analyzed using descriptive statistics. Comparison between groups will be done using t-tests or ANOVA procedures. Other inferential statistical analysis will be conducted as appropriate.
Level of fatty acid synthase by western blot | Up to 72 hours after starting chemotherapy
  Results will be analyzed using descriptive statistics. Comparison between groups will be done using t-tests or ANOVA procedures. Other inferential statistical analysis will be conducted as appropriate.
Number of mononuclear cells per sample determined by cell isolation | Up to 72 hours after starting chemotherapy
  Results will be analyzed using descriptive statistics. Comparison between groups will be done using t-tests or analysis of variance (ANOVA) procedures. Other inferential statistical analysis will be conducted as appropriate.
Oxygen consumption rate | Up to 72 hours after starting chemotherapy
  Results will be analyzed using descriptive statistics. Comparison between groups will be done using t-tests or ANOVA procedures. Other inferential statistical analysis will be conducted as appropriate.
Number of viable samples | Up to 72 hours after starting chemotherapy
  Results will be analyzed using descriptive statistics. Comparison between groups will be done using t-tests or ANOVA procedures. Other inferential statistical analysis will be conducted as appropriate.
Level of hexokinase by western blot | Up to 72 hours after starting chemotherapy
  Results will be analyzed using descriptive statistics. Comparison between groups will be done using t-tests or ANOVA procedures. Other inferential statistical analysis will be conducted as appropriate.
Level of phosphofructokinase-1 by western blot | Up to 72 hours after starting chemotherapy
  Results will be analyzed using descriptive statistics. Comparison between groups will be done using t-tests or ANOVA procedures. Other inferential statistical analysis will be conducted as appropriate.
Level of phosphoglycerate mutase by western blot | Up to 72 hours after starting chemotherapy
  Results will be analyzed using descriptive statistics. Comparison between groups will be done using t-tests or ANOVA procedures. Other inferential statistical analysis will be conducted as appropriate.
Total level of pyruvate kinase M2 by western blot | Up to 72 hours after starting chemotherapy
  Results will be analyzed using descriptive statistics. Comparison between groups will be done using t-tests or ANOVA procedures. Other inferential statistical analysis will be conducted as appropriate.
Level of pyruvate kinase M2 for phospho-T105 by western blot | Up to 72 hours after starting chemotherapy
  Results will be analyzed using descriptive statistics. Comparison between groups will be done using t-tests or ANOVA procedures. Other inferential statistical analysis will be conducted as appropriate.
Level of phosphofructokinase-2 by western blot | Up to 72 hours after starting chemotherapy
  Results will be analyzed using descriptive statistics. Comparison between groups will be done using t-tests or ANOVA procedures. Other inferential statistical analysis will be conducted as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pardee, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States